CLINICAL TRIAL: NCT02423395
Title: Randomized Study of Orphenadrine' in the Treatment of Muscle Cramps in Patients With Cirrhosis
Brief Title: Study of Orphenadrine' in the Treatment of Muscle Cramps in Patients With Cirrhosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Study director, Tanta University
Organization: Tanta University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: muscle cramps in cirrhotics
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Liver Cirrhosis; Muscle Cramps
MeSH Terms: conditions — Liver Cirrhosis; Muscle Cramp | interventions — Orphenadrine; Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Orphenadrine(Norflex) (Experimental): 50 patients will be treated with orphenadrine 100 mg twice daily for 1 month
  Interventions: Drug: orphenadrine
- Placebo (Placebo Comparator): 50 patients will be given placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: orphenadrine — Orphenadrine in muscle cramps in cirrhotic patients
  Other Names: Norflex
  Arms: Orphenadrine(Norflex)
Drug: Placebo — calcium in muscle cramps in cirrhotic patients
  Other Names: calcium
  Arms: Placebo

SUMMARY:
Muscle cramps are common in patients with liver disease and associated with significantly diminished quality of life. Patients with cirrhosis often experience muscle cramps with varied frequency and severity. The exact mechanisms by which they occur remain unclear, although a number of pathophysiological events unique to liver disease may contribute. Clinical studies have identified alterations in 3 areas: nerve function, energy metabolism, and plasma volume/electrolytes (1) Orphenadrine is an anticholinergic drug with prominent central nervous system (CNS) and peripheral actions used to treat painful muscle spasms and other similar conditions. The combination of anticholinergic effects and CNS penetration make orphenadrine useful for pain of all etiologies, including from: radiculopathy, muscles, and headaches. [3,4]

DETAILED DESCRIPTION:
Muscle cramps are common in patients with liver disease and associated with significantly diminished quality of life. Patients with cirrhosis often experience muscle cramps with varied frequency and severity. The exact mechanisms by which they occur remain unclear, although a number of pathophysiological events unique to liver disease may contribute. Clinical studies have identified alterations in 3 areas: nerve function, energy metabolism, and plasma volume/electrolytes [1].

Although a number of mechanisms for cramps in liver disease have been postulated and have been targeted by medical therapies, a clear picture of the causal events has not emerged. Several agents as vitamin E, human albumin, zinc, taurine, eperisone hydrochloride and branched-chain amino acids have shown some benefit in small uncontrolled studies, although large randomized controlled trials are lacking [2].

Orphenadrine is an anticholinergic drug with prominent central nervous system (CNS) and peripheral actions used to treat painful muscle spasms and other similar conditions. The combination of anticholinergic effects and CNS penetration make orphenadrine useful for pain of all etiologies, including from: radiculopathy, muscles, and headaches. [3,4] Orphenadrine is structurally related to diphenhydramine and carries relatively stronger anticholinergic and weaker sedative properties, It is mostly excreted through the kidneys.[5]

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis
* Muscle cramps( ≥3 cramps per week )

Exclusion Criteria:

* • Allergy to orphenadrine

  * Renal impairment
  * Pregnant and lactating women
  * Peripheral vascular disease
  * Peripheral neuropathy
  * Medications as calcium channel blockers, conjugated estrogens and naproxen. Glaucoma Prostatic enlargement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-01; Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of muscle cramps | 3 months
  questionnaire

SECONDARY OUTCOMES:
Quality of life of these patients | 3 months
  questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Asem A Elfert, Professor, Principal Investigator — TUH; Samah Mosaad, Lecturer, Study Chair — TUH; Lobna Aboaly, Professor, Study Chair — TUH; Walaa ElKhalawany, Lecturer, Study Chair — TUH; Sherief Abd-Elsalam, Lecturer, Study Director — TUH
Locations (1):
- Tanta university hospital, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abd-Elsalam S, Ebrahim S, Soliman S, Alkhalawany W, Elfert A, Hawash N, Elkadeem M, Badawi R. Orphenadrine in treatment of muscle cramps in cirrhotic patients: a randomized study. Eur J Gastroenterol Hepatol. 2020 Aug;32(8):1042-1045. doi: 10.1097/MEG.0000000000001622. PMID 31834056